CLINICAL TRIAL: NCT02030717
Title: Randomized Study of Spinal Anesthesia Compared With Traditional Epidural Anesthesia Concerning Peroperative and Postoperative Pain After Open Nephrectomy in Patients With Renal Cell Carcinoma
Acronym: ASA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University Hospital, Umeå (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 151:2010/81099; 2008-001491-77 (EudraCT Number)
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Pre- and Postoperative Analgesia; Spinal Anesthesia; Renal Cell Carcinoma
Keywords: Spinal anesthesia; Epidural anesthesia; Klonidin; renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal anesthesia (Experimental): The drugs used in the spinal injection are: 12 mg bupivacain, 160 ug morfin och klonidin( < 60 years 75 ug, 60 - 85 years old 60 ug and older than 85 years 45 ug)
  Interventions: Drug: klonidin
- Epidural anesthesia (Active Comparator): Epidural anesthesia patients group gets an epidural catheter at level Th 8- 10 with per- and postoperative infusion with a routine mixture of: bupivacain 1 mg/ml, fentanyl 1 ug/ml, and adrenalin 1 ug/ml) until termination.
  Interventions: Drug: epidural anesthesia

INTERVENTIONS:
Drug: klonidin — spinal injection of 12 mg bupivacain,160 ug morfin och klonidin, according to age
  Other Names: Brand name: Duraclon - FDA Apl No (NDA) 020615.
  Arms: Spinal anesthesia
Drug: epidural anesthesia — epidural anesthesia: patients get an continuous infusion of a solution with bupivacain 1 mg/ml, fentanyl 1 ug/ml and adrenalin 1 ug/ml
  Arms: Epidural anesthesia

SUMMARY:
The study aim to study whether spinal anesthesia (using: bupivacain, morfin och klonidin) can be better than epidural anesthesia during and after open surgery for renal cell carcinoma. Per- and postoperative pain after spinal anesthesia with klonidin can be reduced and, thus, shorten the hospital stay and rehabilitation of the patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients in ASA score I - III, planned to be treated with open radical nephrectomy or nephron-sparing surgery having renal cell carcinoma

Exclusion Criteria:

* patients in ASA score IV-V,
* patients with advanced tumour thrombus in vena cava inferior,
* patients with high risk for bleeding
* patients with previous chronic pain symptoms
* patients having drug abuse
* patients having cognitive deficiencies or dementia disease
* patients with any contraindication of either spinal or epidural anesthesia
* patients younger than 18 years and pregnant woman
* patients having a weight less than 45 kg or weight over 120 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
postoperative mobilisation index | within the first 30 days (plus or minus 5 days) after surgery
  Using a number of variables an index of mobilisation has been created; eg pain (10 graded scale), malaise, intravenous substitution, eating in dining room, Walking outside ward room, passage of stool, carrying urinary bladder catheter, can mobilise out of bed without help

SECONDARY OUTCOMES:
time of hospitalization | within the first 15 days after surgery
  time in hospital after surgery until discharge

OTHER OUTCOMES:
Need of rescue analgetics | within the first 15 days after surgery
  the total amount of analgetics used besides the spinal infusion or the epidural infusion used

CONTACTS AND LOCATIONS:
Overall Officials: Borje Ljungberg, MD, PhD, Study Chair — Umea University
Locations (1):
- Umea University Hospital, Umeå, Sweden

REFERENCES:
- [Derived] Thurm M, Hultin M, Johansson G, Dahlin BI, Winso O, Ljungberg B. Spinal anaesthesia with clonidine: pain relief and earlier mobilisation after open nephrectomy - a randomised clinical trial. J Int Med Res. 2022 Sep;50(9):3000605221126883. doi: 10.1177/03000605221126883. PMID 36177827